CLINICAL TRIAL: NCT06073353
Title: Randomized Controlled Trial of a Psychosocial Mobile Application (THRIVE-M) for Patients Living With Multiple Myeloma
Brief Title: Psychosocial Mobile Application (THRIVE-M) for Patients With Multiple Myeloma
Acronym: THRIVE-M
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-332
Record Dates: First submitted 2023-09-02; First posted 2023-10-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is a double-blind single-site randomized efficacy trial of the THRIVE-M App in 120 patients with multiple myeloma. Patients will be recruited from the Massachusetts General Hospital Cancer Center and randomized in a 1:1 fashion, stratified by diagnosis type (newly diagnosed versus maintenance versus relapsed), to assign each participant to either THRIVE-M versus usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE-M (Experimental): Participants will be recruited from the Massachusetts General Hospital Cancer Center and randomized in a 1:1 fashion, stratified by diagnosis type (newly diagnosed versus maintenance versus relapsed), to THRIVE-M versus usual care.
  Participants will use THRIVE-M following a diagnosis of multiple myeloma to learn how to cope with physical symptoms, articulate their needs and navigate relationships, and focus on self-care while living with multiple myeloma using an iPad provided by the study team or the participant's own iPad.
  Questionnaires (in person, over the computer or telephone, or by mail) will be completed by participants at predetermined days per protocol days.
  Interventions: Behavioral: THRIVE-M
- Usual Care (No Intervention): Participants will be recruited from the Massachusetts General Hospital Cancer Center and randomized in a 1:1 fashion, stratified by diagnosis type (newly diagnosed versus maintenance versus relapsed), to THRIVE-M versus usual care.
  Questionnaires (in person, over the computer or telephone, or by mail) will be completed by participants at predetermined days per protocol days.
  Participants in the usual care arm will receive their usual care with the multiple myeloma team, including all routine supportive care resources (e.g., support from social work, psychology, or psychiatry) offered by the multiple myeloma team to all patients diagnosed with multiple myeloma.
  Patients in both the usual care and THRIVE-M group are permitted to use all supportive care services per usual care. We will track referrals to supportive care services in both groups by reviewing the Electronic Health Record (EHR).

INTERVENTIONS:
Behavioral: THRIVE-M — THRIVE-M is a self-administered psychosocial mobile application for patients living with multiple myeloma that includes the following five modules:
  1. Health module - teaching patients about physical symptoms and strategies to cope with physical symptoms
  2. Relationships module - helping patients articulate different support needs and communication styles in navigating relationships
  3. emotions module - helping patients identify connections between thoughts, feelings, and behaviors, as well as helpful states of mind and gratitude
  4. Lifestyle module - helping patients practice skills for saving up energy and using self-care strategies
  5. Reflection module - teaching patients to reflect on their lives, meaningful relationships, and sense of purpose.
  Each module takes about 15-20 minutes to complete and participants will be instructed to complete all modules within an eight-week period.
  Arms: THRIVE-M

SUMMARY:
This clinical trial aims to evaluate whether a psychosocial mobile application (THRIVE-M), is efficacious for improving quality of life, psychological distress, and fatigue in patients living with multiple myeloma compared to usual care.

DETAILED DESCRIPTION:
Multiple myeloma, the second most common hematologic malignancy, can be associated with severe end-organ destruction and life-threatening complications (e.g., kidney failure, infection, anemia) resulting in significant morbidity (e.g., pain syndromes, fatigue). The protracted course and treatment of multiple myeloma is also characterized by physical symptoms that can undermine psychological well-being, functioning, and quality of life across the illness trajectory and care continuum.

Despite the high psychological burden that may accompany life with multiple myeloma, the special mental health workforce needed to adequately address their psychological needs is limited. Hence, mobile application-delivered psychosocial interventions offer an innovative approach to overcome the shortage of psychosocial services to support the unique needs of patients living with multiple myeloma. With no psychosocial mobile application interventions for patients living with multiple myeloma, we developed a patient-centered, population-specific, mobile-application psychosocial intervention, THRIVE-M, tailored to the unique needs of patients living with multiple myeloma. With this study, we will establish the impact of THRIVE-M on patient-reported outcomes compared to usual care.

The study will use validated questionnaires to measure patients' quality of life, psychological distress symptoms, fatigue, and self-management targets like coping, spiritual well-being, and self-efficacy. Study questionnaires will be completed in the hospital or clinic, with an option to also complete them remotely via a secure web link or a mailed paper copy.

Divine Mercy University is funding this research study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 years or older) with one of the following diagnoses:

  1. newly diagnosed multiple myeloma receiving first-line therapy,
  2. multiple myeloma on maintenance therapy, or
  3. relapsed multiple myeloma receiving 2nd or 3rd line therapy
* Ability to comprehend, read, and respond to questions in English

Exclusion Criteria:

- Patients with acute or unstable psychiatric or cognitive conditions that the treating clinicians believe prohibit informed consent or compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life as measured by the Functional Assessment of Cancer Therapy - Multiple Myeloma (FACT-MM) scale | 8 weeks
  Compare quality of life between participants receiving THRIVE-M versus usual care as measured by the Functional Assessment of Cancer Therapy-Multiple Myeloma (FACT-MM) at 8 weeks. the FACT-MM score ranges 0-164 with higher scores indicating better quality of life
  Higher scores on the FACT-MM (range 0-164) indicate better quality of life.

SECONDARY OUTCOMES:
Quality of life longitudinally based on the FACT-MM scale | Up to 15 weeks
  Compare quality of life using the Functional Assessment of Cancer therapy (FACT-MM) between the two groups. The FACT-MM ranges 0-164 with higher scores indicating better quality of life.
  Higher scores on the HADS anxiety subscale (range 0-21) indicate greater anxiety symptoms.
Anxiety Symptoms based on the Hospital Anxiety and Depression Scale | Up to 15 weeks
  Compare anxiety symptoms between participants receiving THRIVE-M versus usual care as measured by the Hospital Anxiety and Depression Scale (HADS)-anxiety subscale. The HADS-Anxiety subscale ranges from 0-21 with higher scores indicating worse anxiety symptoms.
  Higher scores on the HADS anxiety subscale (range 0-21) indicate greater anxiety symptoms.
Depression Symptoms based on the Hospital Anxiety and Depression Scale | Up to 15 weeks
  Compare depression symptoms between participants receiving THRIVE-M versus usual care as measured by the Hospital Anxiety and Depression Scale (HADS)-depression. The HADS-Depression subscale ranges from 0-21 with higher scores indicating worse depression symptoms.
  Higher scores on the HADS-depression subscale (range 0-21) indicate greater depression symptoms.
Post-traumatic Stress Disorder (PTSD) Symptoms based on the PTSD Checkist | Up to 15 weeks
  Compare PTSD symptoms between participants receiving THRIVE-M versus usual care as measured by the PTSD Checklist-Civilian Version. The PTSD checklist score ranges from 17-85 with higher scores indicating worse post-traumatic stress symptoms.
  Higher Scores on the PTSD Checklist-Civilian Version (range 17-85) indicate greater PTSD symptoms.
Fatigue based on the FACT-Fatigue Scale | Up to 15 weeks
  Compare fatigue between participants receiving THRIVE-M versus usual care as measured by the Functional Assessment of Cancer Therapy-Fatigue (FACT-Fatigue). The FACT-Fatigue ranges from 0-52 with higher scores indicating lower fatigue.
  Higher scores on the FACT-Fatigue (range 0-52) indicate worse fatigue.

OTHER OUTCOMES:
Coping based on the Measure of Current Status Part A (MOCS-A) scale | Up to 15 weeks
  Compare coping between participants receiving THRIVE-M versus usual care as measured by the Measure of Current Status Part A (MOCS-A). The MOCS-A ranges from 0-52 with higher scores indicating greater coping skills.
  Higher scores on the MOCS-A (range 0-52) indicate better coping.
Self-efficacy based on the Cancer Self-Efficacy Scale (CASE) | Up to 15 weeks
  Compare self-efficacy between participants receiving THRIVE-M versus usual care as measured by the Cancer self-efficacy Scale (CASE). The Case ranges from 0-170 with higher scores indicating higher self-efficacy.
  Higher scores on the CASE (range 0-170) indicate greater self-efficacy.
Spiritual Well-being based on the FACT-spiritual scale | Up to 15 weeks
  Compare spiritual well-being between participants receiving THRIVE-M versus usual care as measured by the Functional Assessment of Chronic Illness Therapy-Spiritual (FACIT-Sp-12). The FACIT-SP-12 score ranges from 0-48 with higher scores indicating better spiritual wellbeing.
  Higher scores on the FACIT-Sp-12 (range 0-48) indicate greater spiritual well-being.
Optimism based on the Life Orientation Test-Revised (LOT-R) scale | Up to 15 weeks
  Compare optimism between participants receiving THRIVE-M versus usual care as measured by the Life Orientation Test-Revised (LOT-R). The score range is 0-24 with higher scores indicating better optimism
  Higher scores on the LOT-R (range 0-24) indicate greater optimism.
Life Satisfaction based on the Satisfaction with Life Scale (SWLS) | Up to 15 weeks
  Compare life satisfaction between participants receiving THRIVE-M versus usual care as measured by the Satisfaction with Life Scale (SWLS). The SWLS ranges 5-25 with higher scores indicating better life satisfaction.
  Higher scores on the SWLS (range 5-35) indicate greater life satisfaction.
Positive Affect based on the Positive Affect Schedule (PANAS) | Up to 15 weeks
  Compare positive affect between participants receiving THRIVE-M versus usual care as measured by the positive affect subscale of the Positive Affect Schedule (PANAS). The score ranges 10-50, with higher scores indicating more positive affect.
  Higher scores on the positive affect scale of the PANAS (range 10-50) indicate greater positive affect.
Gratitude based on the Gratitude Questionniare-6 | Up to 15 weeks
  Compare gratitude between participants receiving THRIVE-M versus usual care as measured by the Gratitude Questionnaire-6 (GQ-6). the score range 6-42 with higher scores indicating more gratitude.
  Higher scores on the GQ-6 (range 6-42) indicate greater gratitude.
Loneliness based on the Cancer Loneliness Scale (CLS) | Up to 15 weeks
  Compare loneliness between participants receiving THRIVE-M versus usual care as measured by the Cancer Loneliness Scale (CLS). The score ranges 20-80 with higher scores indicating greater feelings of loneliness
  Higher scores on the CLS (range 15-75) indicate greater loneliness.
Usability of THRIVE-M app based on the System Usability Scale | Up to 8 weeks
  We will use the System Usability Scale to assess the usability of THRIVE-M for those receiving the intervention. This scale ranes 0-100 with higher scores indicating better usability.
  Higher scores on the System Usability Scale ( range 0-100) indicate better usability.

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Mass General Brigham innovations team at http://www.partners.org/innovation